CLINICAL TRIAL: NCT06741020
Title: Hepatic Arterial Infusion Chemotherapy and Immunotherapy (HAICI) as Neoadjuvant Treatment for Resectable Hepatocellular Carcinoma in BCLC A/B Stage Beyond Up to Seven Criteria: An Open-Label, Single-Arm, Pilot Study
Brief Title: Hepatic Arterial Infusion Chemotherapy and Immunotherapy for Hepatocellular Carcinoma
Acronym: HAICI
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yuhua Zhang, MD, Prof., Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-413
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Neoadjuvant therapy; Beyond up to seven; Hepatic arterial infusion chemotherapy and immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Intervention Model Description: Patients will receive A combination of Oxaliplatin, Calcium folinate, 5-Fluorouracil and Adebrelimab with transhepatic arterial infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HAICI group (Experimental): Day 1: Adebrelimab 1200mg, administer over 1 hour. Day 1: Oxaliplatin 85mg/m², administer over 1-3 hours; Day 1: Leucovorin calcium 400mg/m², administer over 3-4 hours; Day 1: Fluorouracil 400mg/m², administer as a bolus infusion (50ml/min) at the 4th hour; Fluorouracil 2400mg/m², continue infusion for more than 46 hours; If the patient has two or more supplying arteries, consider placing a perfusion catheter in the main artery for infusion, and use iodinated oil, doxorubicin or idarubicin, oxaliplatin, and other drugs for chemoembolization in other arteries.
  The above treatment regimen is repeated every 3 weeks for a treatment cycle.
  Interventions: Drug: Adebrelimab, Oxaliplatin, Fluorouracil,Leucovorin

INTERVENTIONS:
Drug: Adebrelimab, Oxaliplatin, Fluorouracil,Leucovorin — Chemotherapy drugs including Oxaliplatin, Fluorouracil,Leucovorin and immunotherapy durgs Adebrelimab will infuse to liver by transarterial catheter toward to the lesion.

SUMMARY:
Dear Sir/Madam, We would like to invite you to participate in this clinical research, which has been approved by the Medical Ethics Committee of Zhejiang Cancer Hospital. This informed consent form provides you with detailed information to help you decide whether or not to participate in this study. Please read it carefully, and ensure you fully understand it or get satisfactory answers to your questions before making your decision. If you have any questions, please feel free to consult the researchers, and we will provide you with comprehensive explanations.

Hepatic artery infusion chemotherapy (HAIC) has recently become a popular local treatment method for liver cancer. A large Phase III clinical study from Sun Yat-sen University Cancer Center demonstrated that in a randomized comparison of HAIC versus transarterial chemoembolization (TACE) for unresectable large hepatocellular carcinoma (≥7 cm), the objective response rate (ORR) for HAIC was 46%, while TACE had an ORR of only 18%, with a statistically significant difference between the two. Additionally, HAIC showed advantages over TACE in terms of progression-free survival (PFS) and overall survival (OS), reducing the risk of disease progression by 43% and the risk of death by 42%. In subgroups based on age, sex, performance status, alpha-fetoprotein levels, tumor size, and number of tumors, HAIC consistently demonstrated superior PFS and OS. A study from Taiwan indicated that for patients with advanced liver cancer with portal vein tumor thrombus, the ORR for the HAIC group reached 22.86%, compared to 26.09% for those using immune checkpoint inhibitors alone, and an ORR of 50.00% for the group receiving HAIC combined with immune checkpoint inhibitors.

FOLFOX (fluorouracil, leucovorin, and oxaliplatin) has shown positive results as a systemic treatment regimen for advanced liver cancer, with an ORR of 8.15%, a PFS of 2.93 months, and an OS of 6.47 months in comparative studies. When used as a treatment option in advanced liver cancer through hepatic artery infusion, its ORR increased to 31.5%, PFS to 7.8 months, and OS to 13.9 months.

Common immune checkpoint inhibitors include PD-1 monoclonal antibodies and PD-L1 monoclonal antibodies. PD-1 antibodies prevent immune evasion by blocking PD-1 on immune cells, while PD-L1 antibodies block PD-L1 on tumor cells to inhibit their interaction, thus preventing immune evasion. Therefore, PD-1 monoclonal antibodies primarily target immune cells, while PD-L1 monoclonal antibodies primarily target tumor cells. This leads us to attempt hepatic artery infusion of PD-L1 monoclonal antibodies, utilizing a high-concentration saturation infusion method to maximally block PD-L1 on tumor cells and reduce tumor immune evasion. Concurrently, combining FOLFOX-HAIC localized chemotherapy leads to the release of tumor necrosis antigens, facilitating immune system activity.

Thus, we aim to utilize hepatic artery infusion to deliver both PD-L1 monoclonal antibodies and chemotherapy into the liver, killing tumors with high concentrations of chemotherapy, which will lead to antigen release that aids subsequent immune drug effectiveness while reducing suppressive factors in the immune microenvironment, such as Tregs and M2 macrophages. This approach will help change the inhibitory status of the immune microenvironment and provide a foundation for subsequent immunotherapy.

In BCLC staging, stage A patients and some stage B patients have resectable liver cancer. However, factors affecting tumor staging, such as maximum tumor diameter and tumor quantity, are also considered high-risk recurrence factors in clinical models. Therefore, later tumor staging itself is a high-risk factor for tumor recurrence.

In 2009, Professor Mazzaferro and colleagues proposed the Up-to-Seven criteria (the sum of maximum tumor diameter and tumor number not exceeding 7). Patients who met this criteria and received liver transplantation had a five-year survival rate as high as 71%. Liver cancer patients exceeding the Up-to-Seven criteria are considered unsuitable candidates for liver transplantation, as exceeding this limit indicates a poor tumor biological behavior. Furthermore, the criteria align with the primary surgical treatment staging (CNLC Ia-IIa) recommended in the "Primary Liver Cancer Diagnosis and Treatment Guidelines (2024 Edition)" published by China's National Health Commission. Therefore, we plan to conduct a neoadjuvant study targeting resectable liver cancer exceeding the Up-to-Seven criteria, using hepatic artery chemotherapy combined with immune checkpoint inhibitor (PD-L1 monoclonal antibody) infusion as the treatment regimen.

DETAILED DESCRIPTION:
Overall Design

1. Screening Period For patients willing to participate in this clinical study, an informed consent form (in duplicate, with one copy kept by the researcher and one by the patient) will be signed. The researcher will screen for eligibility based on inclusion and exclusion criteria, with all screening tests to be completed between 28 and 0 days before treatment. Patients who meet the inclusion and exclusion criteria will enter the treatment phase.
2. Neoadjuvant Treatment Period 2.1 Establishment of Arterial Infusion Pathway Interventional radiologists will be responsible for catheter placement through the femoral artery or distal radial artery, with the catheter tip adjusted in real-time under DSA monitoring to the distal end of the hepatic artery (beyond the bifurcation of the gastroduodenal artery).

   2.2 Infusion of Hepatic Artery Chemotherapy Drugs and Immune Checkpoint Inhibitors Day 1: Adebrelimab 1200 mg, infused over 1 hour. Day 1: Oxaliplatin 85 mg/m², infused over 1-3 hours. Day 1: Calcium folinate 400 mg/m², infused over 3-4 hours. Day 1: 5-Fluorouracil 400 mg/m², bolus injection during the 4th hour (50 ml/min); 5-Fluorouracil 2400 mg/m², infused continuously for more than 46 hours. If a patient has two or more feeding arteries, consideration may be given to placing an infusion catheter in the main artery, while other arteries may use iodized oil, doxorubicin, or oxaliplatin for chemotherapy embolization.

   This treatment regimen is repeated every 3 weeks. An evaluation will be conducted at the end of each treatment cycle. Patients who achieve Objective Response Rate (ORR) will proceed to the surgical phase, where the researcher will determine whether to perform laparoscopic minimally invasive or open radical surgery. Patients who do not achieve ORR may undergo up to three additional cycles of treatment. Those who achieve ORR will undergo radical surgery three weeks after stopping the treatment. In cases where patients do not achieve ORR, the researcher will evaluate if radical surgery is feasible. If it is feasible, surgery will be performed three weeks after stopping treatment; if not, the patient will be submitted for multidisciplinary discussion regarding subsequent treatment plans. If surgery is delayed due to drug-related side effects within four weeks after obtaining ORR, it will be recorded as a surgical delay, and the time beyond this point will be noted as the duration of the surgery extension.
3. Perioperative Period Complete preoperative assessments and evaluations will be conducted, with surgery performed using either minimally invasive or open techniques. The method of liver resection may be anatomical or non-anatomical resection.
4. Postoperative Adjuvant Treatment Postoperative adjuvant treatment: Patients who achieve ORR in the neoadjuvant treatment phase will receive intravenous Adebrelimab 1200 mg every three weeks. Patients with postoperative pathological negative Microvascular Invasion (MVI) will continue treatment for six months, while those with positive MVI will continue for twelve months. For patients who did not achieve ORR but underwent surgical treatment, the subsequent adjuvant treatment plan will be discussed by the multidisciplinary team (MDT).
5. Safety Follow-up 5.1 Pre-treatment Safety Follow-up: Ensure that the patient's physical condition is in a generally normal state before treatment. A complete blood count, biochemical tests, coagulation function, and electrocardiogram must be completed within seven days prior to treatment to ensure the patient's condition meets pre-treatment requirements.

   5.2 Post-treatment Safety Follow-up: This follow-up is used to monitor damage to the patient's physical condition after treatment, facilitating early correction of any abnormalities. Blood counts and biochemical tests must be completed within three days after treatment; if there is bone marrow suppression or liver/kidney function damage, correction must be achieved before entering the next treatment phase.

   5.3 Periodic Safety Follow-up: This is to monitor damage caused by the cumulative dose of treatment drugs. Tests will include chest CT, cardiac troponin, cortisol (8 AM), and thyroid function, with re-evaluation every treatment cycle.
6. Survival Follow-up This study is exploratory, with the primary endpoint being Objective Response Rate (ORR). However, the time to recurrence (for patients who underwent surgery after neoadjuvant treatment) and progression-free survival (for patients who did not undergo surgery) will still be recorded for every patient participating in the study, as well as overall survival time.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years;
2. Preoperative pathological diagnosis or clinically diagnosed liver cancer meeting EASL/AASLD diagnostic criteria. No prior systemic chemotherapy, immunotherapy, targeted therapy, or other anti-tumor treatments for HCC;
3. Staging in BCLC Stage A or B, and beyond the Up-to-Seven criteria but deemed resectable (negative margins and remaining liver volume sufficient to meet body needs);
4. ECOG performance status score of 0 before the first medication in the study;
5. Liver function classified as Child-Pugh Class A and ICG retention rate at 15 minutes ≤ 10%;
6. Estimated survival time of at least 6 months;
7. Organ function levels meet the requirements and are capable of tolerating surgery before the first medication in the study; Key organ function indicators must meet the following criteria: Hemoglobin ≥ 90 g/L, Neutrophil count ≥ 1.5 × 10⁹/L, Platelet count ≥ 100 × 10⁹/L; Aspartate or Alanine aminotransferase ≤ 5 times the upper limit of normal (ULN), Alkaline phosphatase ≤ 2.5 ULN, Serum albumin ≥ 30 g/L; Serum creatinine < 1.5 ULN; International Normalized Ratio (INR) ≤ 2 or Prothrombin Time (PT) exceeding the upper limit of normal ≤ 6 seconds; Serum creatinine ≤ 1.5 ULN, Creatinine clearance ≥ 60 mL/min.
8. Male and female participants with reproductive potential must agree to use effective contraception throughout the study period;
9. Sign a consent form agreeing to provide previously stored blood samples, tumor tissue specimens, or fresh biopsy tumor lesions.

Exclusion Criteria:

1. Pathological diagnosis of non-hepatocellular carcinoma;
2. Previous treatment for liver cancer-related chemotherapy, radiotherapy, radiofrequency ablation, interventional therapies and targeted therapy, immunotherapy, or surgical procedures (excluding prior non-tumor-related surgeries or diagnostic biopsies);
3. Preoperative assessment indicates the tumor is unresectable;
4. Viral load limitations: hepatitis B virus (HBV) DNA > 2000 copies/ml, hepatitis C virus (HCV) RNA > 1000;
5. Long-term hormone users require ongoing systemic hormone treatment (equivalent to > 10 mg prednisone/day) or any other form of immunosuppressive therapy;
6. Clinical significant bleeding events or bleeding tendencies within 3 months prior to enrollment or currently receiving thrombolytic or anticoagulant treatment;
7. History of autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis, etc.;
8. Active severe clinical infection (> Grade 2, NCI-CTCAE Version 5.0), including active tuberculosis; history of active tuberculosis infection within the past year without receiving formal anti-tuberculosis treatment or ongoing active tuberculosis; known or suspected active autoimmune diseases;
9. Uncontrolled diabetes (fasting blood glucose ≥ 10 mmol/L), severe lung disease (such as acute lung disease, pulmonary fibrosis affecting lung function, interstitial lung disease. However, resolved radiation pneumonitis is excluded);
10. Clinically significant cardiovascular disease; hypertension that is poorly controlled by antihypertensive medications (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
11. Recipients of renal replacement therapy;
12. History of other malignancies within the last 5 years. However, cured skin basal cell carcinoma or cervical carcinoma in situ is excluded;
13. Other conditions that are expected to render the participant unable to tolerate surgical treatment;
14. Allergic reactions to any components of the study drug;
15. Presence of alcohol dependence, mental illnesses, pregnancy (or breastfeeding), or other conditions that make participation in clinical trials inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 12 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all randomized subjects whose objective response is either a CR or PR.

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | Up to 12 months
  DCR is defined as the percentage of participants who have objective response of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1.
Time to Response (TTR) | From date of first dose of study drug until achieveing objective response.
  The duration between treatment start and achieve partial response or complete response.
Surgery Delay (SD) | Up to 6 months
  If surgery cannot be performed due to drug-related side effects within 4 weeks after obtaining the ORR, it is deemed a surgical delay, and the time exceeding this point will be recorded as the surgical extension time.
Treatment-related adverse events | Up to 12 months
  Safety will be evaluated according to the NCI-CTCAE Version 5.0.

OTHER OUTCOMES:
Pathological response rate (PRR) | 1 month after patients recieved liver resection.
  The proportion of tumor necrosis in patients undergoing surgical treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazzaferro V, Llovet JM, Miceli R, Bhoori S, Schiavo M, Mariani L, Camerini T, Roayaie S, Schwartz ME, Grazi GL, Adam R, Neuhaus P, Salizzoni M, Bruix J, Forner A, De Carlis L, Cillo U, Burroughs AK, Troisi R, Rossi M, Gerunda GE, Lerut J, Belghiti J, Boin I, Gugenheim J, Rochling F, Van Hoek B, Majno P; Metroticket Investigator Study Group. Predicting survival after liver transplantation in patients with hepatocellular carcinoma beyond the Milan criteria: a retrospective, exploratory analysis. Lancet Oncol. 2009 Jan;10(1):35-43. doi: 10.1016/S1470-2045(08)70284-5. Epub 2008 Dec 4. PMID 19058754
- [Background] Yang P, Qiu J, Li J, Wu D, Wan X, Lau WY, Yuan Y, Shen F. Nomograms for Pre- and Postoperative Prediction of Long-term Survival for Patients Who Underwent Hepatectomy for Multiple Hepatocellular Carcinomas. Ann Surg. 2016 Apr;263(4):778-86. doi: 10.1097/SLA.0000000000001339. PMID 26135698
- [Background] Shen L, Qi H, Chen S, Cao F, Xie L, Wu Y, Ma W, Song Z, Yuan H, Zhang T, Li D, Wen X, Chen Q, Li W, Zhang X, Fan W. Cryoablation combined with transarterial infusion of pembrolizumab (CATAP) for liver metastases of melanoma: an ambispective, proof-of-concept cohort study. Cancer Immunol Immunother. 2020 Sep;69(9):1713-1724. doi: 10.1007/s00262-020-02566-z. Epub 2020 Apr 24. PMID 32333081
- [Background] Lyu N, Wang X, Li JB, Lai JF, Chen QF, Li SL, Deng HJ, He M, Mu LW, Zhao M. Arterial Chemotherapy of Oxaliplatin Plus Fluorouracil Versus Sorafenib in Advanced Hepatocellular Carcinoma: A Biomolecular Exploratory, Randomized, Phase III Trial (FOHAIC-1). J Clin Oncol. 2022 Feb 10;40(5):468-480. doi: 10.1200/JCO.21.01963. Epub 2021 Dec 14. PMID 34905388
- [Background] Wu JS, Hong TC, Wu HT, Lin YJ, Chang TT, Wang CT, Liu WC, Hsieh MT, Wu IC, Chen PJ, Chen CY, Lin SH, Chuang CH, Han MZ, Chen HP, Tsai HM, Kuo HY. Hepatic arterial infusion chemotherapy and immune checkpoint inhibitors, alone or in combination, in advanced hepatocellular carcinoma with macrovascular invasion: a single-centre experience in Taiwan. J Gastrointest Oncol. 2023 Apr 29;14(2):849-862. doi: 10.21037/jgo-22-858. Epub 2023 Apr 10. PMID 37201085
- [Background] Li QJ, He MK, Chen HW, Fang WQ, Zhou YM, Xu L, Wei W, Zhang YJ, Guo Y, Guo RP, Chen MS, Shi M. Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin Versus Transarterial Chemoembolization for Large Hepatocellular Carcinoma: A Randomized Phase III Trial. J Clin Oncol. 2022 Jan 10;40(2):150-160. doi: 10.1200/JCO.21.00608. Epub 2021 Oct 14. PMID 34648352
- [Background] Xia Y, Tang W, Qian X, Li X, Cheng F, Wang K, Zhang F, Zhang C, Li D, Song J, Zhang H, Zhao J, Yao A, Wu X, Wu C, Ji G, Liu X, Zhu F, Qin L, Xiao X, Deng Z, Kong X, Li S, Yu Y, Xi W, Deng W, Qi C, Liu H, Pu L, Wang P, Wang X. Efficacy and safety of camrelizumab plus apatinib during the perioperative period in resectable hepatocellular carcinoma: a single-arm, open label, phase II clinical trial. J Immunother Cancer. 2022 Apr;10(4):e004656. doi: 10.1136/jitc-2022-004656. PMID 35379737
- [Background] Marron TU, Fiel MI, Hamon P, Fiaschi N, Kim E, Ward SC, Zhao Z, Kim J, Kennedy P, Gunasekaran G, Tabrizian P, Doroshow D, Legg M, Hammad A, Magen A, Kamphorst AO, Shareef M, Gupta NT, Deering R, Wang W, Wang F, Thanigaimani P, Mani J, Troncoso L, Tabachnikova A, Chang C, Akturk G, Buckup M, Hamel S, Ioannou G, Hennequin C, Jamal H, Brown H, Bonaccorso A, Labow D, Sarpel U, Rosenbloom T, Sung MW, Kou B, Li S, Jankovic V, James N, Hamon SC, Cheung HK, Sims JS, Miller E, Bhardwaj N, Thurston G, Lowy I, Gnjatic S, Taouli B, Schwartz ME, Merad M. Neoadjuvant cemiplimab for resectable hepatocellular carcinoma: a single-arm, open-label, phase 2 trial. Lancet Gastroenterol Hepatol. 2022 Mar;7(3):219-229. doi: 10.1016/S2468-1253(21)00385-X. Epub 2022 Jan 20. PMID 35065058
- [Background] Zhou WP, Lai EC, Li AJ, Fu SY, Zhou JP, Pan ZY, Lau WY, Wu MC. A prospective, randomized, controlled trial of preoperative transarterial chemoembolization for resectable large hepatocellular carcinoma. Ann Surg. 2009 Feb;249(2):195-202. doi: 10.1097/SLA.0b013e3181961c16. PMID 19212170
- [Background] Gosavi R, Chia C, Michael M, Heriot AG, Warrier SK, Kong JC. Neoadjuvant chemotherapy in locally advanced colon cancer: a systematic review and meta-analysis. Int J Colorectal Dis. 2021 Oct;36(10):2063-2070. doi: 10.1007/s00384-021-03945-3. Epub 2021 May 4. PMID 33945007
- [Background] De Lena M, Zucali R, Viganotti G, Valagussa P, Bonadonna G. Combined chemotherapy-radiotherapy approach in locally advanced (T3b-T4) breast cancer. Cancer Chemother Pharmacol. 1978;1(1):53-9. doi: 10.1007/BF00253147. PMID 373908
- [Background] Xia YX, Zhang F, Li XC, Kong LB, Zhang H, Li DH, Cheng F, Pu LY, Zhang CY, Qian XF, Wang P, Wang K, Wu ZS, Lyu L, Rao JH, Wu XF, Yao AH, Shao WY, Fan Y, You W, Dai XZ, Qin JJ, Li MY, Zhu Q, Wang XH. [Surgical treatment of primary liver cancer:a report of 10 966 cases]. Zhonghua Wai Ke Za Zhi. 2021 Jan 1;59(1):6-17. doi: 10.3760/cma.j.cn112139-20201110-00791. Chinese. PMID 33412628
- [Background] Zeng H, Chen W, Zheng R, Zhang S, Ji JS, Zou X, Xia C, Sun K, Yang Z, Li H, Wang N, Han R, Liu S, Li H, Mu H, He Y, Xu Y, Fu Z, Zhou Y, Jiang J, Yang Y, Chen J, Wei K, Fan D, Wang J, Fu F, Zhao D, Song G, Chen J, Jiang C, Zhou X, Gu X, Jin F, Li Q, Li Y, Wu T, Yan C, Dong J, Hua Z, Baade P, Bray F, Jemal A, Yu XQ, He J. Changing cancer survival in China during 2003-15: a pooled analysis of 17 population-based cancer registries. Lancet Glob Health. 2018 May;6(5):e555-e567. doi: 10.1016/S2214-109X(18)30127-X. PMID 29653628